CLINICAL TRIAL: NCT05064839
Title: Imaging for the Evaluation of Transthyretin Cardiac Amyloidosis Prevalence of Patients Over 65 Hospitalized in Cardiology Wards (the IMPACT Study)
Acronym: IMPACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A00732-39
Record Dates: First submitted 2021-08-26; First posted 2021-10-01 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Transthyretin Cardiac Amyloidosis
Keywords: cardiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bony scintigraphy (Experimental): Bony scintigraphy within 1 to 4 months after inclusion
  Interventions: Procedure: Bony scintigraphy

INTERVENTIONS:
Procedure: Bony scintigraphy — Bony scintigraphy (99mTc-Hydromethylene diphosphonate) will be performed in all patients with hypertrophy of the left ventricle

SUMMARY:
Heart failure with preserved ejection and hypertrophic cardiomyopathy are common diseases and often associated with transthyretin cardiac amyloidosis (TTR-CM), especially in elderly people. Nevertheless, research of TTR-CM is recommended in patients with ventricular hypertrophy without other cause such as valvular disease or hypertension. Therefore, the exact prevalence of TTR-CM remains unknown. We aim to determine the prevalence of TTR-CM in patients with ventricular hypertrophy and aged ≥ 60 years old, hospitalized in our cardiology department (CHU de Poitiers) by performing bone scintigraphy and research of AL amyloidosis.

DETAILED DESCRIPTION:
Not Provided

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 60 years, hospitalised in cardiology wards of the Centre Hospitalier Universitaire of Poitiers
* Left ventricle hypertrophy on echocardiography
* Patient able to comply with study procedures
* Patient legally free and not subject to any custody, guardianship, tutelage or subordination measures
* Patient having signed an informed consent after clear and fair information on the study

Exclusion Criteria:

* CardiacTransplant
* Complex congenital cardiopathies
* Know diagnosis of amylosis
* Contra-indication to bony scintigraphy : hypersensitivity to sodium oxidronate or one of its excipients, or to one of the components of radiopharmaceutic marked product ;
* Subject not able to comply with study procedures
* Patients not benefiting from a Social Security scheme or not benefiting from it through a third party
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, patients staying in a health or social establishment, adults under legal protection, and patients in emergency situation.
* Women not menopausal

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a positive bone scintigraphy (perugini score> or = 2) in the absence of AL cardiac amyloidosis. | At Visit 2, one to four months after inclusion visit.
  Percentage of patients with a positive bone scintigraphy (perugini score> or = 2) in the absence of AL cardiac amyloidosis in patients over 60 years hospitalised in cardiology wards, with an hypertrophy of the left ventricle on transthoracic echocardiography (thickness of the left ventricle at the end of diastole >12mm), whatever the possible cause of hypertrophy of the left ventricle (other potential cause not excluded), and without prior diagnosis of cardiac amylosis.

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. de Poitiers, Poitiers, France